CLINICAL TRIAL: NCT06856577
Title: A Multi-Center, Randomized, Double-Masked, Active-Comparator-Controlled, Phase 3 Study to Evaluate the Efficacy and Safety of Ixoberogene Soroparvovec (Ixo-vec) in Participants With Neovascular Age-Related Macular Degeneration (ARTEMIS)
Brief Title: Efficacy and Safety Study of Ixoberogene Soroparvovec (Ixo-vec) in Participants With Neovascular Age-Related Macular Degeneration
Acronym: ARTEMIS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Adverum Biotechnologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ADVM-022-12
Record Dates: First submitted 2025-02-26; First posted 2025-03-04 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Neovascular Age-Related Macular Degeneration (nAMD); Wet AMD
Keywords: Ixoberogene soroparvovec; Ixo-vec; Aflibercept; Neovascular age-related macular degeneration; nAMD; ADVM; ADVM-022; ADVM-022-12; Wet AMD; wAMD; Wet Age-related Macular Degeneration; CNV; Neovascular AMD; AAV; AAV vector; AAV.7m8-aflibercept; AAV.7m8; Gene therapy; Eye disease; Blindness; Adeno-associated viruses
MeSH Terms: conditions — Eye Diseases; Blindness | interventions — aflibercept

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ixo-vec (Experimental): Participants will receive 3 monthly loading doses of aflibercept 2 mg IVT, a single IVT injection of Ixo-vec 6 x 10^10 vg/eye at Week 1, and sham injections every 8 weeks
  Interventions: Genetic: Ixo-vec; Drug: Aflibercept
- Aflibercept (Active Comparator): Participants will receive 3 monthly loading doses of aflibercept 2 mg IVT, a sham injection at Week 1, and aflibercept 2 mg IVT every 8 weeks.
  Interventions: Drug: Aflibercept

INTERVENTIONS:
Genetic: Ixo-vec — Ixo-vec will be administered intravitreally.
  Arms: Ixo-vec
Drug: Aflibercept — Aflibercept will be administered intravitreally.

SUMMARY:
This is a multi-center, randomized, double-masked, active-comparator-controlled, Phase 3 study in a broad participant population (treatment-naïve and treatment-experienced) with neovascular (wet) age-related macular degeneration (nAMD). The study will evaluate a single intravitreal (IVT) injection of Ixo-vec compared to an active comparator. The primary endpoint of this study is the mean change in best corrected visual acuity (BCVA) of Ixo-vec compared to an active comparator measured at an average of Weeks 52 and 56.

Safety, tolerability, and efficacy will be evaluated throughout the study.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the non-inferiority in efficacy of a single intravitreal (IVT) injection of Ixo-vec 6 x 10^10 vector genome (vg)/eye compared to an active comparator.

Neovascular or wet age-related macular degeneration (nAMD) is a degenerative ocular disease associated with the infiltration of abnormal blood vessels in the retina from the underlying choroid layer and is a leading cause of blindness in patients over 65 years of age. The abnormal angiogenic process in nAMD is stimulated and modulated by vascular endothelial growth factor (VEGF). Treatment of nAMD requires frequent intravitreal (IVT) injections of VEGF inhibitors (anti-VEGF) administered every 4-16 weeks. Ixo-vec (also known as ADVM-022 or AAV.7m8-aflibercept) is a gene therapy product being developed for the treatment of nAMD. Ixo-vec is designed to reduce the current treatment burden which often results in undertreatment and vision loss in patients with nAMD receiving anti-VEGF therapy in clinical practice.

Safety, tolerability, and efficacy will be evaluated throughout this study. The primary endpoint of this study is the mean change in best corrected visual acuity (BCVA) of Ixo-vec compared to an active comparator measured at an average of Weeks 52 and 56 post-treatment.

Due to the long duration of the Screening period, this study will be considered fully enrolled when randomization has been completed.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide informed consent (or have a legally authorized representative who is able and willing to provide informed consent) prior to any study assessments and procedures and comply with the study requirements and visits.
2. Male or female with a diagnosis of CNV secondary to nAMD in the study eye, with nAMD disease activity at Screening Visit 1.
3. At least 50 years old at Screening Visit 1.
4. An Early Treatment Diabetic Retinopathy Study (ETDRS) BCVA letter score of 35 - 78 (approximate Snellen equivalent of 20/200 to 20/32) in the study eye at Screening Visit 1.
5. Demonstrated a meaningful anatomic response to anti-VEGF therapy during screening
6. Able to reliably use eye drops per protocol

Exclusion Criteria:

General Exclusion Criteria

1. History of a medical condition giving reasonable suspicion of a condition that contraindicates the use of Ixo-vec, compromises the participant's ability to comply with the planned study activities, or that might affect the interpretation of the results of the study or render the participant at high risk for treatment complications in the opinion of the Investigator. History of severe coronavirus disease (COVID-19) infection may meet this exclusion criteria if, in the opinion of the Investigator, it is likely to lead to any important complications.
2. Received any prior gene therapy.
3. Prior treatment with any non-gene therapy investigational medicinal product (IMP) or medical device in the study eye within 3 months of Screening Visit 1 or 5 half-lives of the IMP prior to dosing with Ixo-vec, whichever is longer.
4. Female participants who are pregnant or breastfeeding or who intend to become pregnant or breastfeed in the future.
5. History or evidence of any of the following cardiovascular diseases:

   1. Myocardial infarction in the 6-month period prior to Week 1.
   2. Uncontrolled hypertension defined as systolic blood pressure > 160 mmHg or diastolic blood pressure > 100 mmHg during screening.
   3. Stroke in the 6-month period prior to Week 1.
6. History of ongoing bleeding disorders. The use of aspirin or other anticoagulants (e.g., Factor Xa inhibitors) is permitted.
7. Use of systemic immunosuppressive drugs within 90 days prior to Screening Visit 1. Short courses of oral corticosteroids are permitted, as well as any inhaled, intra-articular, nasal or dermal steroid use.
8. Evidence of poorly controlled diabetes or glycated hemoglobin (HbA1c) ≥ 8.0% during screening

Ocular Exclusion Criteria

1. Any active ocular or periocular infection in the study eye from Screening Visit 1.
2. History or evidence of the following in the study eye:

   1. Intraocular or refractive surgery within 5 months prior to Week 1.
   2. Any previous penetrating keratoplasty or vitrectomy.
   3. Any previous panretinal photocoagulation.
   4. Any previous submacular surgery, other surgical intervention (including port delivery system) or laser treatment for age related macular degeneration.
3. Any history or evidence of retinal detachment (with or without repair) or retinal pigment epithelium rip/tear in the study eye, as determined by the Investigator during screening or at Week 1.
4. Uncontrolled ocular hypertension or glaucoma in the study eye from Screening Visit 1 to Week 1 or current use of ≥ 2 IOP lowering medications or normal tension glaucoma/suspect in the study eye or history of any of the following procedures in the study eye prior to Week 1:

   * Incisional glaucoma surgery (i.e., glaucoma drainage implant/shunt or trabeculectomy)
   * Ocular angle-based surgery (i.e., goniotomy or canaloplasty)
   * Minimally Invasive Glaucoma Surgery (MIGS) in the study eye.
   * Angle-based glaucoma surgery (e.g., Argon or Selective Laser Trabeculoplasty)
5. Any history of intraocular pressure (IOP) elevation related to topical steroid administration in either eye.
6. Any history of uveitis or inflammation (grade trace or above) except mild anticipated post operative inflammation that resolved in either eye.
7. Any history of treatment with complement inhibitors for geographic atrophy in the study eye.
8. Known history of ocular herpes simplex virus, varicella-zoster virus, or cytomegalovirus, including viral uveitis, retinitis, or keratitis in either eye.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2026-12-22 (Estimated); Study Completion 2030-11-23 (Estimated)

PRIMARY OUTCOMES:
Mean change from Baseline in Best-Corrected Visual Acuity (BCVA) based on an average at Weeks 52 and 56 | Baseline, Week 52 and Week 56
  BCVA will be measured using an Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity chart.

SECONDARY OUTCOMES:
Mean number of aflibercept IVT injections received | Week 4 through Week 56
Percentage of participants with worsened BCVA | Through Week 56
  BCVA measured by ETDRS
Percentage of participants with improved BCVA | Through Week 56
  BCVA measured by ETDRS
Mean change from Baseline in BCVA over time based on an average at Weeks 52 and 56 | Through Week 56
  BCVA measured by ETDRS
Mean change from Week 1 in BCVA based on an average at Weeks 52 and 56 | Week 1 through Week 56
  BCVA measured by ETDRS
Percentage of participants with BCVA of 73 letters or more from Week 4 through Week 56 | Week 4 through Week 56
Mean change in Central Subfield Thickness (CST) from Baseline over time through Week 56 | Through Week 56
  CST as measured by spectral domain optical coherence tomography (SD-OCT)
Percentage of participants with CST ≤ 300 μm over time through Week 56 | Through Week 56
  CST will be assessed by a CRC using SD-OCT
Mean number of CST fluctuations > 50 μm from Week 1 over time through Week 56 | Week 1 through Week 56
  CST will be assessed by a CRC using SD-OCT images and the mean number of fluctuations with thickness of more than 50 μm will be summarized
Percentage of participants with CST fluctuations > 50 μm from Week 1 over time through Week 56 | Week 1 through Week 56
  CST will be assessed using SD-OCT
Percent reduction in mean rate of annualized anti-Vascular Endothelial Growth Factor (VEGF) injections | Through Week 56
  Percent reduction in mean rate of annualized anti-VEGF injections will be assessed relative to the reduction in mean rate of annualized anti-VEGF injections received in the year prior to screening in treatment-experienced participants
Percentage of participants who were aflibercept injection-free | Week 4 through Week 56
Percentage of participants who received 0 or 1 aflibercept injection | Week 4 through Week 56
Mean change in area of Choroidal Neovascularization (CNV) lesion from Baseline over time through Week 56 | Baseline through Week 56
  CNV is the infiltration of abnormal blood vessels in the retina from the underlying choroid layer. It will be assessed by a CRC using SD-OCT.
Mean change in macular volume from Baseline over time through Week 56 | Baseline through Week 56
  Macular volume will be measured as part of the full ophthalmic examination.
Percentage of participants without Intraretinal Fluid (IRF) over time through Week 56 | Through Week 56
  IRF will be assessed using SD-OCT
Percentage of participants without Subretinal Fluid (SRF) over time through Week 56 | Through Week 56
  SRF will be assessed using SD-OCT
Percentage of participants without IRF and/or SRF over time through Week 56 | Through Week 56
  IRF and SRF will be assessed using SD-OCT
Time to dry retina | Through Week 56
  Dry retina is defined as no IRF or SRF (i.e., absence of either). IRF and SRF will be assessed using SD-OCT
Time to sustained dry retina | Through Week 56
  Sustained dry retina is defined as no IRF or SRF (i.e., absence of either) maintained for 2 consecutive visits.
Number of participants who experienced ocular adverse events | Through Week 56
  The number of participants who experience an ocular adverse event will be summarized.
Number of participants who experienced mild, moderate or severe ocular adverse events | Through Week 56
  The number of participants who experience a mild, moderate or severe ocular adverse event will be summarized.
Number of participants who experienced non-ocular adverse events | Through Week 56
  The number of participants who experience a non-ocular adverse event will be summarized.
Number of participants who experienced mild, moderate or severe non-ocular adverse events | Through Week 56
  The number of participants who experience a mild, moderate or severe non-ocular adverse event will be summarized.
Mean change in 25-item National Eye Institute Visual Function Questionnaire (NEI VFQ-25) total and subscale scores | Day 1 to Week 28 and Week 56
  The NEI VFQ-25 measures vision-targeted patient-reported outcomes of individuals with chronic eye diseases. It comprises 25 questions. The assessment generates an overall composite score and includes the following subscales: global vision rating, difficulty with near vision activities, difficulty with distance vision activities, limitations in social functioning due to vision, role limitations due to vision, dependency on others due to vision, mental health symptoms due to vision, driving difficulties, limitations with peripheral and color vision, and ocular pain. A decrease in the NEI VFQ-25 score represents an improvement in disease severity.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Turpcu, PhD, Study Director — Adverum Biotechnologies, Inc.
Locations (79):
- United States (79):
  - Adverum Clinical Site 223, Gilbert, Arizona
  - Adverum Clinical Site 178, Phoenix, Arizona
  - Adverum Clinical Site 126, Phoenix, Arizona
  - Adverum Clinical Site 229, Scottsdale, Arizona
  - Adverum Clinical Site 159, Tucson, Arizona
  - Adverum Clinical Site 198, Springdale, Arkansas
  - Adverum Clinical Site 109, Bakersfield, California
  - Adverum Clinical Site 100, Beverly Hills, California
  - Adverum Clinical Site 201, Campbell, California
  - Adverum Clinical Site 172, Encino, California
  - Adverum Clinical Site 169, Fullerton, California
  - Adverum Clinical Site 224, Huntington Beach, California
  - Adverum Clinical Site 215, Redlands, California
  - Adverum Clinical Site 164, Riverside, California
  - Adverum Clinical Site 140, Sacramento, California
  - Adverum Clinical Site 212, Sacramento, California
  - Adverum Clinical Site 175, Santa Barbara, California
  - Adverum Clinical Site 202, Torrance, California
  - Adverum Clinical Site 189, Walnut Creek, California
  - Adverum Clinical Site 200, Denver, Colorado
  - Adverum Clinical Site 116, Lakewood, Colorado
  - Adverum Clinical Site 165, Waterford, Connecticut
  - Adverum Clinical Site 184, Deerfield Beach, Florida
  - Adverum Clinical Site 176, Fort Lauderdale, Florida
  - Adverum Clinical Site 221, Fort Myers, Florida
  - Adverum Clinical Site 236, Gainesville, Florida
  - Adverum Clinical Site 168, Jacksonville, Florida
  - Adverum Clinical Site 214, Lakeland, Florida
  - Adverum Clinical Site 213, Orlando, Florida
  - Adverum Clinical Site 230, Pensacola, Florida
  - Adverum Clinical Site 124, Pompano Beach, Florida
  - Adverum Clinical Site 183, South Miami, Florida
  - Adverum Clinical Site 120, St. Petersburg, Florida
  - Adverum Clinical Site 193, Tampa, Florida
  - Adverum Clinical Site 182, Augusta, Georgia
  - Adverum Clinical Site 149, ‘Aiea, Hawaii
  - Adverum Clinical Site 179, Oak Forest, Illinois
  - Adverum Clinical Site 207, Oak Park, Illinois
  - Adverum Clinical Site 195, Carmel, Indiana
  - Adverum Clinical Site 205, Carmel, Indiana
  - Adverum Clinical Site 197, Hagerstown, Maryland
  - Adverum Clinical Site 204, Hagerstown, Maryland
  - Adverum Clinical Site 167, Detroit, Michigan
  - Adverum Clinical Site 216, Madison, Mississippi
  - Adverum Clinical Site 163, Southaven, Mississippi
  - Adverum Clinical Site 190, St Louis, Missouri
  - Adverum Clinical Site 171, Teaneck, New Jersey
  - Adverum Clinical Site 225, Liverpool, New York
  - Adverum Clinical Site 196, Asheville, North Carolina
  - Adverum Clinical Site 234, Cary, North Carolina
  - Adverum Clinical Site 186, Durham, North Carolina
  - Adverum Clinical Site 211, Greensboro, North Carolina
  - Adverum Clinical Site 220, Hickory, North Carolina
  - Adverum Clinical Site 209, Wake Forest, North Carolina
  - Adverum Clinical Site 219, Winston-Salem, North Carolina
  - Adverum Clinical Site 181, Erie, Pennsylvania
  - Adverum Clinical Site 110, Philadelphia, Pennsylvania
  - Adverum Clinical Site 208, Charleston, South Carolina
  - Adverum Clinical Site 222, Ladson, South Carolina
  - Adverum Clinical Site 122, West Columbia, South Carolina
  - Adverum Clinical Site 144, Rapid City, South Dakota
  - Adverum Clinical Site 123, Abilene, Texas
  - Adverum Clinical Site 127, Austin, Texas
  - Adverum Clinical Site 108, Bellaire, Texas
  - Adverum Clinical Site 227, Burleson, Texas
  - Adverum Clinical Site 194, Dallas, Texas
  - Adverum Clinical Site 188, Houston, Texas
  - Adverum Clinical Site 218, Katy, Texas
  - Adverum Clinical Site 162, McAllen, Texas
  - Adverum Clinical Site 151, San Antonio, Texas
  - Adverum Clinical Site 185, San Antonio, Texas
  - Adverum Clinical Site 232, San Marcos, Texas
  - Adverum Clinical Site 228, Schertz, Texas
  - Adverum Clinical Site 107, The Woodlands, Texas
  - Adverum Clinical Site 231, The Woodlands, Texas
  - Adverum Clinical Site 199, Lynchburg, Virginia
  - Adverum Clinical Site 131, Spokane, Washington
  - Adverum Clinical Site 152, Morgantown, West Virginia
  - Adverum Clinical Site 187, Wausau, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Adverum is committed to transparency. Appropriately de-identified participant-level datasets and supporting documents may be shared under proper conditions (e.g. when contractually permitted to do so and when participants provide appropriate consent). Individual patient-level data sets would only be shared following completion of this study (and any associated studies), completion of all applicable regulatory submissions and consistent with any regulatory rules or laws, and criteria established by Adverum, our collaborators and/or industry best practices. Data-sets and/or documents may be modified (eg, de-identified) or redacted to protect participant identity and to protect sensitive or confidential information. For inquiries, please contact us at datasharing@adverum.com.